CLINICAL TRIAL: NCT00324012
Title: Phase II Trial With Taxotere and Cisplatin in Non-operable Adrenocortical Carcinoma
Brief Title: Trial With Taxotere and Cisplatin in Non-operable Adrenocortical Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gedske Daugaard, Associate professor, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02 262098
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenocortical Carcinoma; cisplatin; taxotere
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): taxotere and cisplatin day one every three weeks
  Interventions: Drug: cisplatin, taxotere

INTERVENTIONS:
Drug: cisplatin, taxotere — cisplatin 75 mg/m2 Taxotere 75 mg/m2
  Other Names: docetaxel

SUMMARY:
The trial is a phase II trial in adrenocortical carcinoma (ACC), a rare malignancy with poor prognosis. It will provide results leading to the establishment of the effect of the included drugs. The regimen consists of cisplatin plus taxotere. Over a period of 1-2 years this national trial will include 19-36 patients with advanced ACC from different centres in Denmark. Patients not responding to the first line treatment will be switched to the alternative regimen. The primary objective of this trial is to investigate response rate. Secondary endpoints are survival, time to progression, best overall response rate and duration of response.

DETAILED DESCRIPTION:
Treatment every three weeks, evaluation after 2 cycles, CTC criterias used for toxicity evaluation

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adrenocortical carcinoma
* Locally advanced or metastatic disease not amenable to radical surgery resection (Stage III-IV)
* Radiologically measurable disease
* ECOG performance status 0-2
* Life expectancy > 3 months
* Age ≥18 years
* Adequate bone marrow reserve (neutrophils > 1500/mm3 and platelets > 100,000/mm3)
* Effective contraception in pre-menopausal female and male patients
* Patient's written informed consent
* Ability to comply with the protocol procedures (including availability for follow-up visits)
* Previous palliative surgery, radiotherapy or radiofrequency ablation is acceptable as long as radiologically monitorable disease is verifiable afterwards.

Exclusion Criteria:

* History of prior malignancy, except for cured non-melanoma skin cancer, curatively in situ cervical carcinoma, or other cancers treated with no evidence of disease for at least five years.
* Previous cytotoxic chemotherapy for adrenocortical carcinoma
* Renal insufficiency (serum creatinine ≥2 mg/dl or creatinine clearance ≤ 60 ml/min)
* Hepatic insufficiency (serum bilirubin ≥2 x the institutional upper limit of normal range and/or serum transaminases ≥ 3 x the institutional upper limit of normal range; exception: in patients on mitotane, transaminase levels up to 5 x the institutional upper limit of normal range are acceptable)
* Pregnancy or breast feeding
* Known hypersensitivity to any drug included in the treatment protocol
* Presence of active infection
* Any other severe clinical condition that in the judgment of the local investigator would place the patient at undue risk or interfere with the study completion
* Current treatment with other experimental drugs and/or previous participation in clinical trials with other experimental agents for adrenocortical carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
response rate | in months

SECONDARY OUTCOMES:
Survival, time to progression, best overall response rate and duration of response | survival at 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gedske Daugaard, M.D., DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Oncology 5073, Rigshospitalet, Copenhagen, Denmark